CLINICAL TRIAL: NCT03014128
Title: Musculoskeletal Pathologies of the Upper Extremity in Surgical Device Mechanics
Acronym: PEIN
Status: Completed | Type: Observational
Sponsor: District Hospital, Tuttlingen (Other)
Responsible Party: Sponsor
Other Study IDs: PEIN-78532
Record Dates: First submitted 2016-12-20; First posted 2017-01-09 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: musculoskeletal disorders; upper extremity; work; surgical instruments
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Inspection and Packaging: self-descriptive
  Interventions: Other: Clinical examination and data processing of questionnaires
- Grinding, Polishing and Matting: self-descriptive
  Interventions: Other: Clinical examination and data processing of questionnaires
- All other employees at Aesculap (not in first 2 groups): including administration and offices as well as all other mechanical workplaces
  Interventions: Other: Clinical examination and data processing of questionnaires

INTERVENTIONS:
Other: Clinical examination and data processing of questionnaires — xy

SUMMARY:
Work-related upper extremity musculoskeletal disorders (WRUEMSDs) have shown to be related to many occupational situations and specific industries. However, there is conflicting information about monotonous and repetitive activities. In this context, the profession of surgical device mechanics has not been analyzed so far.

The objective of this study is to examine surgical device mechanics at different workplaces with varying work contents and to compare them with a control group without the repetitive workload exposition as described above. The headquarters and main production site of Aesculap are located in Tuttlingen/Germany. Aesculap is the world leading manufacturer of surgical devices.

After statistical power analysis, the investigators plan to randomize and include a total of 90 voluntary test persons in 3 groups (30 persons each). The study will include standardized questionnaires and a physical examination as well as an industry test (Purdue Pegboard Test).

Primary and secondary endpoints were defined to show if significant difference between surgical device mechanics and a control group is present.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* work ability without absence > 2 weeks within the last 3 months
* >5 years on workplace or similar workplace when in group of surgical device mechanics

Exclusion Criteria:

* spinal syndrome in history
* chronic shoulder pain in history
* congenital malformation of the upper extremity/hand
* rheumatoid arthritis or fibromyalgia in history
* actual hand therapy as conservative therapy or therapy after operation due to upper extremity musculoskeletal pathology
* previous operation(s) due to nerve entrapment syndrome or chronic musculoskeletal pathology of the upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees of the Aesculap AG, world leader in production of surgical devices
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder and Hand) Score (questionnaire) | 6 months
  Validated questionnaire for upper extremity assessment (link in the reference section)

SECONDARY OUTCOMES:
Range of wrist motion | 6 months
  wrist extension/flexion, supination/pronation, ulnar/radial abduction (in degrees)
Grip force of the hand | 6 months
  Hydraulic Hand Dynamometer (in kgs)
Finger sensibility | 6 months
  2-Point-Discrimination (in mm)
Stenosing tenosynovitis | 6 months
  Clinical test, focussing on areas of pain, smoothness of finger motion, evidence of locking (= trigger finger) and presence of lump in the palm (0=negative/no pathology, 1=positive/pathology)
De Quervain tenosynovitis | 6 months
  Clinical test, focussing on pain on thumb and wrist movement, focal tenderness and swelling over radial styloid, positive Finkelstein test (pain on passive ulnar deviation) and triggering or crepitus (0=negative/no pathology, 1=positive/pathology)
Nerve entrapment syndromes | 6 months
  Hoffmann's sign: tingling sensation triggered by a mechanical stimulus in the distal part of entrapped nerves (0=negative/no pathology, 1=positive/pathology)
Carpal tunnel syndrome | 6 months
  Phalen maneuver: the test person is asked to hold the wrist in complete and forced flexion for 60 seconds. This provokes symptoms characteristic for carpal tunnel syndrome such as burning, tingling or numb sensation over the thumb, index, middle and ring fingers (0=negative/no pathology, 1=positive/pathology)
Tennis elbow (lateral epicondylitis) | 6 months
  Maudsley's test (= middle finger test): the examiner resists extension of the 3rd digit of the hand, stressing the extensor digitorum muscle and tendon, while palpating the test person's lateral epicondyle (0=negative/no pathology, 1=positive/pathology)
Purdue Pegboard Test | 6 months
  Standardized industrial test to examine uni- and bimanual skill (number of repetitions, point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Lotter, MD, Principal Investigator — Klinikum Landkreis TUT, Zeppelinstraße 21, 78532Tuttlingen/Germany
Locations (1):
- Aesculap AG, Tuttlingen, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Information about the "Disabilities of the Arm, Shoulder and Hand Score (DASH)" — http://www.dash.iwh.on.ca/about-dash